CLINICAL TRIAL: NCT05302011
Title: A Prospective, Single-armed Study to Evaluate the Efficacy and Safety of Neoadjuvant Pembrolizumab Plus Chemotherapy in Resectable Locally Advanced Esophageal Squamous Cell Carcinoma Patients
Brief Title: Neoadjuvant Pembrolizumab Plus Chemotherapy for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Keypoint-1
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — pembrolizumab; Carboplatin; Cisplatin; Drug Therapy; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Pembrolizumab Plus Chemotherapy (Experimental): Neoadjuvant Pembrolizumab Plus Chemotherapy
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin or Cisplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg i.v. day 1-22-43-64
Drug: Carboplatin or Cisplatin — Carboplatin Area Under the Curve(AUC) = 4-5 i.v. day 1-22-43-64 or Cisplatin 75mg/m2 i.v. day 1-22-43-64
  Other Names: chemotherapy
Drug: Docetaxel — 75mg/m2 i.v. day 1-22-43-64
  Other Names: chemotherapy

SUMMARY:
This is a study to evaluate the efficacy and safety of neoadjuvant pembrolizumab plus chemotherapy in resectable locally advanced esophageal squamous cell carcinoma patients

DETAILED DESCRIPTION:
The primary objective of the study is to assess the tumor response (by irRECIST) and pathological response of neoadjuvant pembrolizumab plus chemotherapy (carboplatin, paclitaxel).

Secondary objectives are:

To assess completion of neoadjuvant pembrolizumab plus chemotherapy. To assess toxicities of neoadjuvant pembrolizumab plus chemotherapy To assess completion of neoadjuvant pembrolizumab plus chemotherapy. To assess withdrawal rate from surgery. To assess delay rate from surgery. To assess R0 resection rate. To assess post-operative complications. Progression Free Survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the esophagus.
* Surgical resectable (T3 or T4b, N0 or N+, M0), as determined by Endoscopic Ultra Sound (EUS),Positron Emission Tomography/Computed Tomography (PET/CT), Esophageal MRI and enhanced CT scan of neck, thorax and abdomen.
* Tumor length longitudinal ≤ 10 cm; if larger than 10 cm, inclusion should be discussed with the principal investigator.
* 18≤Age.
* Tumor does not involve gastro-esophageal junction.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematological, renal and hepatic functions defined as:

neutrophiles ≥ 1.5 x 109/L platelets ≥ 100 x 109/L alanine transaminase≤2 x upper normal limit hemoglobin ≥ 5.6 mmol total bilirubin ≤ 1.5 x upper normal limit creatinine clearance (Cockcroft) ≥60 ml/min

* Written, voluntary informed consent

Exclusion Criteria:

* Past or current history of malignancy other than entry diagnosis interfering with prognosis of esophageal cancer.
* T1, T2 tumors or in situ carcinoma.
* metastatic oesophageal cancer.
* Pregnancy (positive serum pregnancy test), planning to become pregnant, and lactation.
* Previous chemotherapy, radiotherapy, and/or treatment with checkpoint inhibitors.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) precluding major surgery.
* Pulmonary fibrosis and/or severely impaired lung function precluding major surgery.
* Pre-existing motor or sensory neurotoxicity greater than World Health Organization (WHO) grade 1.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (>10 mg/day prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent
* Serious underlying medical condition which would impair the ability of the patient to receive the planned treatment, including prior allergic reactions to drugs containing Cremophor, such as teniposide or cyclosporine.
* Has an active infection requiring systemic therapy which has not resolved 3 days (simple infection such as cystitis) to 7 days (severe infection such as pyelonephritis) prior to the first dose of trial treatment.
* Has a diagnosis of acute or chronic hepatitis B, hepatitis C, known immunodeficiency or human immunodeficiency virus (HIV).
* Patients with prior allogeneic stem cell or solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
tumor response | up to 12 months
  assess the tumor response (by irRECIST) of neoadjuvant pembrolizumab plus chemotherapy
pathological response | up to 12 months
  assess the pathological responses (by College of American Pathologists(CAP) classification) of neoadjuvant pembrolizumab plus chemotherapy

SECONDARY OUTCOMES:
Percentage completion of treatment | up to 3 months
  Percentage completion of treatment in neoadjuvant pembrolizumab plus chemotherapy
Incidence and severity of toxicity | up to 12 months
  Incidence and severity of toxicity defined to CTCAE v4.03 and Radiation Oncology Group (RTOG) criteria
Percentage withdrawal rate from surgery | up to 3 months
  Percentage withdrawal rate from surgery due to neoadjuvant related complications
Percentage delay of surgery | up to 3 months
  Percentage delay of surgery due to neoadjuvant related complications
R0 resection rate | up to 3 months
  R0 resection rate
Incidence and severity of post-operative complications to the Clavien-Dindo classification | up to 3 months
  Incidence and severity of post-operative complications to the Clavien-Dindo classification
Disease free survival | up to 24 months
  Disease free survival
Overall survival | up to 24 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China